CLINICAL TRIAL: NCT02533297
Title: Developing Standards for Skill Performance Times in Nursing Clinical Education Program According to Learning Curve
Brief Title: Developing Standards Skill According to the Learning Curves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyedreza Mazloum, Head of Centre ٍvidence- based Research, Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 88490
Record Dates: First submitted 2015-08-14; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Nursing Student
Keywords: standardization,; performance clinical skills; nursing; learning curve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clinical education (Experimental): the researcher used the checklist to assess the student's mastery level skill l while changing a skill and recorded his score on the learning curve based on a 1 (no mastery) to 100 (complete mastery) scoring scale. This procedure continued until the learning curve reached to a plateau state, i.e. either reaching to the full mastery score (100) or revealing no significant change in three subsequent sessions. All the students achieved mastery (the plateau state) after performing the task for at most ten times.
  Interventions: Other: Providing clinical skills conditions

INTERVENTIONS:
Other: Providing clinical skills conditions

SUMMARY:
The aim of the current study was to develop a criterion in terms of the number of sessions required to achieve mastery in DCS based on the learning curve assessment in real clinical situation.

ELIGIBILITY:
Inclusion Criteria:

* Nursing and midwifery students in Mashhad.
* Before the relevant skills in teaching nursing for the theoretical and practical training
* Employment as student work , etc., is not nursing .

Exclusion Criteria:

* Skills into the clinical environment is not done , or a maximum of three times ( contact skills intravenous line , dry dressing , intramuscular injection ) has done .

Defects or diseases that cause skills to do independent problem , no . ( At the discretion of the instructor )

No sign student proficiency , skills required in this section or elsewhere has done .

Student of psychological ( lack of acute stress , etc.) is ready to perform skills . ( At the discretion of the instructor )

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
level of expertise nursing student | in training course (4month follow up)
  The checklist contained steps for performance skill rated on a 1 to 3 scoring scale (1= The researcher used the checklist to assess the student's mastery level while changing a skill and recorded his score on the learning curve based on a 0 (no mastery) to 100 (complete mastery) scoring scale.Required Standard frequency for skills performance based on learning curve plateau, achievement of 75% of expertise and, 75 percent of students who achieved 75% of expertise in the following skills.

REFERENCES:
- [Result] Miri K, Malekzade J, Davoudi N, Mazloum S. How many Times of Intramuscular Injec-tion and Intravenous Catheter Insertion is Essential for Learning? Developing Standards according to the Learning Curves. Iranian Journal of Medical Education. 2013; 13 (6) :457-469